CLINICAL TRIAL: NCT02434120
Title: Validation, for Orbital Tumors, of the MRI Perfusion Curves Typology Established for Salivary Tumors
Brief Title: MRI Perfusion Curves Typology and Orbital Tumors (PERFORM)
Acronym: PERFORM
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ALR_2015_13
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Orbital Tumor
Keywords: MRI; Orbital neoplasm
MeSH Terms: conditions — Orbital Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Orbital masses develop at the expense of the orbital structures lacrimal glands, oculomotor muscles, optic nerve, meningeal spaces, peripheral nerves, bone wall, orbital fat, lymphoid structures or vascular structures. These masses can be tumors, benign or malignant, or pseudotumor, mainly represented by specific or non-specific orbital inflammation.

Pathology is of considerable importance for the diagnosis and the treatment of those masses. However, biopsy or surgical resection of the orbital masses is sometimes difficult and dangerous outside expert centers.

The identification of a non-invasive technique for distinguishing tumors from pseudotumors, thus avoid in some cases a biopsy, would be a major contribution for the patients.

For salivary glands, MRI allows to identify 4 different types of MRI characteristics, one (type C) being related to malignant tumors.

In this study, the investigators will try to see if extrapolation of those data to orbiltal tumors is feasible.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or more
* with orbital mass for which a biopsy and/or a surgical removal is planned
* undergoing an MRI
* before surgery

Exclusion Criteria:

* contra-indication to MRI
* intolerance to constrast agent
* pregnancy
* breast feeding
* patient under a legal protection procedure
* patient denying to participate to the study
* lack of affiliation to a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a MRI because of an orbital mass
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Concordance of the MRI type and the pathological findings as assessed by the kappa coefficient | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation A De Rothschild, Paris, France

REFERENCES:
- [Result] O'Shaughnessy E, Cossec CL, Mambour N, Lecoeuvre A, Savatovsky J, Zmuda M, Duron L, Lecler A. Diagnostic Performance of Dynamic Contrast-Enhanced 3T MR Imaging for Characterization of Orbital Lesions: Validation in a Large Prospective Study. AJNR Am J Neuroradiol. 2024 Mar 7;45(3):342-350. doi: 10.3174/ajnr.A8131. PMID 38453407
- [Result] O'Shaughnessy E, Senicourt L, Mambour N, Savatovsky J, Duron L, Lecler A. Toward Precision Diagnosis: Machine Learning in Identifying Malignant Orbital Tumors With Multiparametric 3 T MRI. Invest Radiol. 2024 Oct 1;59(10):737-745. doi: 10.1097/RLI.0000000000001076. Epub 2024 Apr 11. PMID 38597586